CLINICAL TRIAL: NCT04782934
Title: Early Feasibility and First in Human Study of the YANG System for Continuous Monitoring of Glucose, Ketones and Lactate - The GLOW Study
Brief Title: The GLOW Study - The YANG System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indigo Diabetes NV (Industry)
Collaborators: University Hospital, Antwerp (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: IND007
Record Dates: First submitted 2021-02-24; First posted 2021-03-04 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-03

CONDITIONS: Diabetes Mellitus; Glucose
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- YANG system group (Experimental)
  Interventions: Device: The YANG SENSOR is an active implantable device, for Real Time Continuous Glucose, Lactate and Ketone Measurement

INTERVENTIONS:
Device: The YANG SENSOR is an active implantable device, for Real Time Continuous Glucose, Lactate and Ketone Measurement — The YANG SENSOR is an active implantable device, that is intended to be implanted in the subcutaneous abdominal tissue, approximately 10mm below the skin. The SENSOR is battery powered. The battery is wirelessly recharged through the skin by the YANGEXD, using a charging coil ('Donut') applied to the skin with an adhesive patch at the level of the SENSOR. The 'Donut' also receives data from the sensor.

SUMMARY:
This is an open label, interventional, monocentric, prospective early feasibility study, designed to evaluate the safety of implant and short-term integration into the tissue of the YANG sensor. In addition, the set up will enable data collection which will be used to develop the software algorithm to allow real-time, continuous measurement of glucose, ketone and lactate levels in the interstitial fluid in adults with diabetes mellitus, in a future version of the device.

ELIGIBILITY:
Inclusion Criteria:

T1DM patients

* Subjects willing to sign an informed consent form (ICF),
* Adult subjects, age ≥ 18, ≤ 50 years old
* Body Mass Index (BMI) 20≥, ≤ 27.5 [kg/m2]
* Subjects willing to comply to study protocol requirements (exercises, ketone ester drinks, alcohol, study visits, blood sampling etc)
* Patients with type 1 diabetes mellitus (T1DM) according to WHO criteria, diagnosed for at least 12 months prior to screening
* Subjects being on insulin pump for at least 12 months

Healthy Volunteers

* Subjects willing to sign an informed consent form (ICF),
* Adult subjects, age ≥ 18, ≤ 50 years old
* BMI 20≥, ≤ 27.5
* Subjects willing to comply to study protocol requirements (exercises, ketone ester drinks, alcohol, study visits, blood sampling etc)
* Healthy subjects, as self-declared and confirmed by screening assessments and Principal Investigator's judgment

Exclusion Criteria:

* Subjects with a contraindication to undergo challenging tests (i.e., ischemic heart disease, epilepsy, panhypopituitarism, hypoadrenalism, hypothyroidism, known allergic reaction to ibuprofen/paracetamol/acetylsalicylic acid)
* For people with diabetes: History of severe hypoglycaemia in the previous 6 months. Severe hypoglycaemia is defined as hypoglycaemia resulting in loss of consciousness or seizure
* For people with diabetes: History of diabetic ketoacidosis requiring emergency room visit or hospitalization in the previous 6 months
* Any blood disorder identified by haematocrit <30% or >55%
* History of hepatitis B, hepatitis C, or HIV
* A condition requiring or likely to require magnetic resonance imaging (MRI) during the study duration
* Female subjects who are pregnant, planning on becoming pregnant or nursing
* Any disorder, which in the investigator's opinion might jeopardise subject's safety or compliance with the protocol.
* Coagulation disorder, wound healing and bleeding disorder or taking anticoagulant medication
* Any long-term drug treatments other than insulin, such as statins, low-dose aspirin, fibrates etc.
* The presence of any other active implanted device except for insulin pumps (as defined further in protocol)
* The presence of any other CGM sensor or transmitter located in abdomen (other location is acceptable)
* Impaired fasting glucose or impaired glucose tolerance (for healthy volunteers)
* Any contraindication to the use of the Yang system as listed in the device IFU (i.e. any known allergy to PDMS)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2021-02-25 (Actual); Primary Completion 2021-06-19 (Actual); Study Completion 2021-06-19 (Actual)

PRIMARY OUTCOMES:
Incidence of device-related or sensor insertion/removal procedure-related adverse events | 57 days
Assessment of foreign body reaction due subcutaneous implantation with biopsy | 27 days
  Assessment of i.e. inflammation, infection, tissue vascularization, formation of fibrotic scar tissue
Incidence of sensor failure | 27 days

SECONDARY OUTCOMES:
Collection of users feedback in the form of clinical questionnaire to assess the 'easiness' of surgical procedure with questionnaire | 1 day
Requirements of duration of implantation and explantation procedure | 27 days
Post explantation follow-up | 30 days
  Removal of sutures and wound healing after 10 days post explantation of the sensor. Follow-up via phone call after 30 days

OTHER OUTCOMES:
Assessment of sensor ability to measure glucose and β-hydroxybutyrate and lactate levels to allow the development of the algorithm | 27 days
  Exploratory endpoint
Assessment of influence of interference substances (i.e. ethanol, lactate, ketones, paracetamol, acetylsalicylic acid, sorbitol, fructose, aspartame, ibuprofen, caffeine and ascorbic acid [Vitamin C]) | 27 days
  Exploratory endpoint: blood samples will be taken each 2.5 or 5 min to measure glucose, lactate and ketones. Glucose will also be measured with a CGM. The influence of the confounders on the glucose measurement by the sensor in the interstitial fluid will be investigated.

CONTACTS AND LOCATIONS:
Overall Officials: Christophe De Block, Prof. Dr., Principal Investigator — University Hospital, Antwerp
Locations (1):
- University Hospital Antwerp, Edegem, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] De Ridder F, Braspenning R, Ordonez JS, Klarenbeek G, Lauwers P, Ledeganck KJ, Delbeke D, De Block C. Early feasibility study with an implantable near-infrared spectroscopy sensor for glucose, ketones, lactate and ethanol. PLoS One. 2024 May 3;19(5):e0301041. doi: 10.1371/journal.pone.0301041. eCollection 2024. PMID 38701088